CLINICAL TRIAL: NCT00570843
Title: Phase 4 Masked Comparison of a New PEG Based Artificial Tear and Optive for Comfort, Vision & Wear Time in Patients Wearing Contact Lenses
Brief Title: Masked Comparison of a New PEG Based Artificial Tear and Optive for Comfort, Vision & Wear Time in Patients Wearing Contact Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Christopher Starr, MD, Weill Cornell Medical College- The New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0710009485
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Comfort, Vision and Wear Time

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1. (Active Comparator)
  Interventions: Drug: New PEG based artificial tear
- 2. (Placebo Comparator)
  Interventions: Drug: Optive

INTERVENTIONS:
Drug: New PEG based artificial tear — 1, 2, (in the eye) Instill one drop in the left eye or right eye four times daily (can be used more frequently if needed)
  Arms: 1.
Drug: Optive — 1, 2, (in the eye) Instill one drop in the left eye or right eye four times daily (can be used more frequently if needed)
  Arms: 2.

SUMMARY:
The objective of this study is to evaluate the effect of a new PEG based artificial tear as compared to Optive on comfort, wear time, and vision in patients wearing contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Use of soft contact lenses (e.g. silicone hydrogel lenses, daily disposables etc.) and multipurpose solution for cleaning, including enzyme-based cleaners (ClearCare etc.)
* Able to wear contact lenses for approximately 10-12 hours/day
* Willingness to complete entire length of trial and comply with subjective questionnaire.

Exclusion Criteria:

* Patients taking topical cyclosporine (Restasis)
* Patients currently using Optive for dryness relief.
* Patients wearing hard or rigid gas permeable lenses
* Patients with uncontrolled systemic disease which may confound the results of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Comfort | 1 month

SECONDARY OUTCOMES:
vision and wear time | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Chris Starr, MD, Principal Investigator — The New York Presbyterian Hospital Weill Cornell Medical College
Locations (1):
- The New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York, United States